CLINICAL TRIAL: NCT04570995
Title: Effect of Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA) on Brain Executive Function in Student Athletes
Brief Title: Effect of Fish Oil on Athlete's Executive Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor unable to send smaller necessary capsules
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00068607
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2020-09

CONDITIONS: Brain Health; Brain Function; Brain Development
Keywords: Polyunsaturated fatty Acids; Executive Function abilities
MeSH Terms: interventions — Fish Oils; Eicosapentaenoic Acid; Docosahexaenoic Acids; Safflower Oil; Fatty Acids, Monounsaturated

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, two-arm intervention study
Who Masked: Participant, Investigator
Masking Description: The capsules are of nearly identical color rendering them indistinguishable in appearance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fish oil (Active Comparator): participants will be asked to consume a daily (5 days per week) dietary supplement containing fish oil encapsulated in soft gel capsules.
  Interventions: Dietary Supplement: Fish Oil
- safflower oil (Placebo Comparator): participants will be asked to consume a daily (5 days per week) dietary supplement containing a placebo oil product (safflower oil) encapsulated in soft gel capsules.
  Interventions: Dietary Supplement: Safflower Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — Dietary supplement containing fish oil, encapsulated in soft gel capsules, given 5 days per week
  Other Names: eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)
  Arms: fish oil
Dietary Supplement: Safflower Oil — Dietary supplement containing a placebo oil product (safflower oil), encapsulated in soft gel capsules, given 5 days per week
  Other Names: high oleic acid (18:1, monounsaturated fatty acid)
  Arms: safflower oil

SUMMARY:
The goal of this study is to determine the impact of long chain omega-3 PUFA (Polyunsaturated fatty acids) supplementation on executive function in collegiate athletes in a randomized, double-blind, placebo-controlled trial

DETAILED DESCRIPTION:
The main objective of this study is to determine the effect of daily oral intake of a fish oil capsule enriched in eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) on brain EF (Executive Function) and blood-based biomarkers among male collegiate baseball student athletes over the course of an academic school year

ELIGIBILITY:
Inclusion Criteria:

* Wake Forest University National Collegiate Athletic Association (NCAA) Division I baseball male student athletes cleared to participate in university athletics as determined by the team physician
* Age >/=18 years

Exclusion Criteria:

* Unwillingness to consume a daily dietary supplement over the course of the study
* Allergy to dietary supplement components
* Lipid-lowering medication use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Barkley Deficits in Executive Functioning Scale (BDEFS) | visit #2 (~6-8 weeks after baseline)
  Evaluate dimensions of adult executive functioning in daily life - self administered - Items are answered on a 4-point scale ranging from "1= Never or rarely" to " 4 = Very often"; α's range from 0.91 to 0.96. Higher scores are interpreted as indicating greater deficits in EF - The Barkley Deficits in Executive Functioning Scale is an 89 item self-report measure of executive functioning.
Stroop Test | visit #2 (~6-8 weeks after baseline)
  Subjects will be asked to read words of colors, state the colors of various letters to test processing speed, and state the color of the font of a word when the actual word describes a conflicting color to test response inhibition (executive functioning).
  Three scores, as well as an interference score, are generated using the number of items completed on each page, with higher scores reflecting better performance and less interference on reading ability. T-Scores of 40 or less are considered "low." Word, color, and color-word T-Scores above 40 or are considered "normal".
Stroop Test | Baseline, Day 1
  Subjects will be asked to read words of colors, state the colors of various letters to test processing speed, and state the color of the font of a word when the actual word describes a conflicting color to test response inhibition (executive functioning).
  Three scores, as well as an interference score, are generated using the number of items completed on each page, with higher scores reflecting better performance and less interference on reading ability. T-Scores of 40 or less are considered "low." Word, color, and color-word T-Scores above 40 or are considered "normal".
Trail Making Test | visit #2 (~6-8 weeks after baseline)
  Visual attention, task switching - self administered - The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.
  The test results are reported as the time that took to complete. Longer times denotes worse outcomes.
Trail Making Test | Baseline, Day 1
  Visual attention, task switching - self administered - The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.
  The test results are reported as the time that took to complete. Longer times denotes worse outcomes.
Stop-Signal Test | visit #2 (~6-8 weeks after baseline)
  Response inhibition - self administered - stop signal task is a test of inhibition of prepotent responses. It requires the participant to respond as quickly as possible to a predetermined stimulus, the go trial, but to abort any response when a subsequently presented stop signal is displayed.
  Speed and accuracy on the go trials are measured. The stop signal reaction time is calculated and reported
Stop-Signal Test | Baseline, Day 1
  Response inhibition - self administered - stop signal task is a test of inhibition of prepotent responses. It requires the participant to respond as quickly as possible to a predetermined stimulus, the go trial, but to abort any response when a subsequently presented stop signal is displayed.
  Speed and accuracy on the go trials are measured. The stop signal reaction time is calculated and reported
Digit Span | visit #2 (~6-8 weeks after baseline)
  Working memory - self administered -Digit Span measures verbal short-term memory, defined as the system that allows for temporary storage of information, and is crucial in everyday tasks such as remembering a telephone number or understanding long sentences - The average digit span for normal adults without error is seven plus or minus two. The Digit Span test is a measure of verbal short-term/working memory. Scores range from 0 to 28, with higher scores indicating better verbal short-term/working memory.
Digit Span | Baseline, Day 1
  Working memory - self administered -Digit Span measures verbal short-term memory, defined as the system that allows for temporary storage of information, and is crucial in everyday tasks such as remembering a telephone number or understanding long sentences - The average digit span for normal adults without error is seven plus or minus two. The Digit Span test is a measure of verbal short-term/working memory. Scores range from 0 to 28, with higher scores indicating better verbal short-term/working memory.
Wisconsin Card Sort Test | visit #2 (~6-8 weeks after baseline)
  Will be administered to assess preservation and abstract thinking. The The task measures how well people can adapt to the changing rules, and their cognitive flexibility.
  The number of perseverative errors in Wisconsin Card Sorting Task is the most robust variable of the task to assess cognitive flexibility. Higher scores show an impairment of cognitive flexibility.
Wisconsin Card Sort Test | Baseline, Day 1
  Will be administered to assess preservation and abstract thinking. The The task measures how well people can adapt to the changing rules, and their cognitive flexibility.
  The number of perseverative errors in Wisconsin Card Sorting Task is the most robust variable of the task to assess cognitive flexibility. Higher scores show an impairment of cognitive flexibility.
Circulating levels of fatty acids - EPA (eicosapentaenoic acid) in plasma | visit #2 (~6-8 weeks after baseline)
  centrifuged to isolate plasma for EPA fatty acid analysis
Circulating levels of fatty acids - EPA on red blood cells | visit #2 (~6-8 weeks after baseline)
  centrifuged to isolate red blood cells for EPA fatty acid analysis
Circulating levels of fatty acids - DHA (docosahexaenoic acid) on Red blood cells | visit #2 (~6-8 weeks after baseline)
  centrifuged to isolate red blood cells for DHA fatty acid analysis
Circulating levels of fatty acids - DHA in plasma | visit #2 (~6-8 weeks after baseline)
  centrifuged to isolate plasma for DHA fatty acid analysis

SECONDARY OUTCOMES:
Capsule consumption compliance | Visits 2 (Week~6-8 weeks after baseline ) and visit 5 (up to 9 months)
  Percentage capsules taken
Weight | Visits 1 to 5, from baseline up to 9 months
BMI | Visits 1 to 5, from baseline up to 9 months
Waist circumference | Visits 1 to 5, from baseline up to 9 months
Hip circumferences | Visits 1 to 5, from baseline up to 9 months
Depression, Anxiety and Stress Scale (DASS) | Visits 1 to 5, from baseline up to 9 months
  Designed to measure the negative emotional states of depression, anxiety and stress - It consists of three 14-item subscales with each item scored on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Total scores are calculated by summing the items on each subscale, giving a score range of 0-42 on each subscale. Scores above 20, 14 and 25 on the depression, anxiety and stress subscales respectively are indicative of severe levels. Higher scores denotes worse outcomes.
Inflammatory and/or injury biomarkers (e.g., isoprostanes) | Visits 1 to 5, from baseline up to 9 months
  quantify plasma levels of inflammatory biomarker assays
Levels of inflammatory and/or injury biomarkers (creatinine kinase) | Visits 1 to 5, from baseline up to 9 months
Levels of inflammatory and/or injury biomarkers (ROS) (Reactive oxygen species) | Visits 1 to 5, from baseline up to 9 months
  quantify plasma levels of inflammatory biomarker assays
Levels of Inflammatory and/or injury biomarkers (IGF) (Insulin-like growth factor 1) | Visits 1 to 5, from baseline up to 9 months
  quantify plasma levels of inflammatory biomarker assays
Levels of inflammatory and/or injury biomarkers (TNF) (Tumor necrosis factor) | Visits 1 to 5, from baseline up to 9 months
  quantify plasma levels of inflammatory biomarker assays
Levels of inflammatory and/or injury biomarkers (CRP) (C-reactive protein) | Visits 1 to 5, from baseline up to 9 months
  quantify plasma levels of inflammatory biomarker assays
Levels of inflammatory biomarkers (IL-6, IL-8, IL-10) (Interleukin) | Post study - 9 months
  quantify plasma levels of inflammatory biomarker assays
Sleep patterns | 4 Visits during 9 months (approximately 6-8 week intervals)
  Time spent in each sleep stage: Light, REM, Slow Wave (Deep), and Awake.
Reaction time assessment | weekly intervals for 9 months of study
  Baseball performance, assessed by reaction time assessment using the DynaVision system
Heart rate variability | From baseline up to 9 months
Heart rate | From baseline up to 9 months
Respiratory rate | From baseline up to 9 months
Barkley Deficits in Executive Functioning Scale (BDEFS) | From Visit 3 (week ~12-16 weeks after baseline) to visit 5 (up to 9 months)
  Evaluate dimensions of adult executive functioning in daily life - self administered - Items are answered on a 4-point scale ranging from "1= Never or rarely" to " 4 = Very often"; α's range from 0.91 to 0.96. Higher scores are interpreted as indicating greater deficits in EF - The Barkley Deficits in Executive Functioning Scale is an 89 item self-report measure of executive functioning.
Stroop Test | From Visit 3 (week ~12-16 weeks after baseline) to visit 5 (up to 9 months)
  Subjects will be asked to read words of colors, state the colors of various letters to test processing speed, and state the color of the font of a word when the actual word describes a conflicting color to test response inhibition (executive functioning).
  Three scores, as well as an interference score, are generated using the number of items completed on each page, with higher scores reflecting better performance and less interference on reading ability. T-Scores of 40 or less are considered "low." Word, color, and color-word T-Scores above 40 or are considered "normal".
Trail Making Test | From Visit 3 (week ~12-16 weeks after baseline) to visit 5 (up to 9 months)
  Visual attention, task switching - self administered - The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.
  The test results are reported as the time that took to complete. Longer times denotes worse outcomes.
Stop-Signal Test | From Visit 3 (week ~12-16 weeks after baseline) to visit 5 (up to 9 months)
  Response inhibition - self administered - stop signal task is a test of inhibition of prepotent responses. It requires the participant to respond as quickly as possible to a predetermined stimulus, the go trial, but to abort any response when a subsequently presented stop signal is displayed.
  Speed and accuracy on the go trials are measured. The stop signal reaction time is calculated and reported
Digit Span | From Visit 3 (week ~12-16 weeks after baseline) to visit 5 (up to 9 months)
  Working memory - self administered -Digit Span measures verbal short-term memory, defined as the system that allows for temporary storage of information, and is crucial in everyday tasks such as remembering a telephone number or understanding long sentences - The average digit span for normal adults without error is seven plus or minus two. The Digit Span test is a measure of verbal short-term/working memory. Scores range from 0 to 28, with higher scores indicating better verbal short-term/working memory.
Wisconsin Card Sort Test | From Visit 3 (week ~12-16 weeks after baseline) to visit 5 (up to 9 months)
  Will be administered to assess preservation and abstract thinking. The The task measures how well people can adapt to the changing rules, and their cognitive flexibility.
  The number of perseverative errors in Wisconsin Card Sorting Task is the most robust variable of the task to assess cognitive flexibility. Higher scores show an impairment of cognitive flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Elaheh Rahbar, PhD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Innis SM. Dietary omega 3 fatty acids and the developing brain. Brain Res. 2008 Oct 27;1237:35-43. doi: 10.1016/j.brainres.2008.08.078. Epub 2008 Sep 9. PMID 18789910
- [Background] McNamara RK, Able J, Jandacek R, Rider T, Tso P, Eliassen JC, Alfieri D, Weber W, Jarvis K, DelBello MP, Strakowski SM, Adler CM. Docosahexaenoic acid supplementation increases prefrontal cortex activation during sustained attention in healthy boys: a placebo-controlled, dose-ranging, functional magnetic resonance imaging study. Am J Clin Nutr. 2010 Apr;91(4):1060-7. doi: 10.3945/ajcn.2009.28549. Epub 2010 Feb 3. PMID 20130094
- [Background] Vesco AT, Young AS, Arnold LE, Fristad MA. Omega-3 supplementation associated with improved parent-rated executive function in youth with mood disorders: secondary analyses of the omega 3 and therapy (OATS) trials. J Child Psychol Psychiatry. 2018 Jun;59(6):628-636. doi: 10.1111/jcpp.12830. Epub 2017 Oct 24. PMID 29063592

DOCUMENTS (1):
  • Informed Consent Form (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04570995/ICF_000.pdf